CLINICAL TRIAL: NCT04162184
Title: Increasing Linkage to Family Planning Care for Individuals With Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deborah Rinehart, Research Scientist, Denver Health and Hospital Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-2621; 1 FPRPA006064-01-00 (Other Grant/Funding Number: HHS Office of Population Affairs)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Family Planning Services; Substance-Related Disorders; Opiate Substitution Treatment; Sexual Health
Keywords: family planning; opioid use disorder; patient navigation; reproductive health; sexual health; substance use disorder; health education
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Health Education | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Educator Intervention (Other): As the population of focus in this study is diverse, including men and women regardless of pregnancy desire, the primary focus for the intervention for this study will be education, particularly for men. All participants that enroll in the study will be offered the intervention. The study health educator will use the PATH (Parenthood/Pregnancy Attitude, Timing, and How) framework questions to initially guide the conversation. Depending on the participant's desires, the educator will provide education on other topics such as sexually transmitted infections (STIs) and we will also navigate to clinical services as needed. The health educator will use a study manual to guide all intervention activities including engagement. Additionally, the health educator will collect data on intervention outreach, engagement, topics discussed, participant needs and outcomes.
  Interventions: Behavioral: Sexual Health Initiative for Navigation and Education (SHINE) Health Educator Intervention

INTERVENTIONS:
Behavioral: Sexual Health Initiative for Navigation and Education (SHINE) Health Educator Intervention — a brief health educator-led behavioral intervention focused on educating, identifying reproductive health needs, and linking to services if desired
  Other Names: SHINE Intervention

SUMMARY:
This study will utilize mixed methods to develop and assess the feasibility and acceptability of a health educator intervention designed to connect patients in recovery from substance use disorder to reproductive health education and services.

DETAILED DESCRIPTION:
Developing effective reproductive health interventions for individuals in treatment for substance use disorder is an important public health priority. In the US nearly half (45%) of all pregnancies are unplanned and studies have consistently found this rate to be much higher among individuals in substance treatment, almost 90%. There is a paucity of research on interventions to support the family planning care of this population. The primary goal of this project is to identify an innovative delivery model to address the family planning needs of individuals of reproductive age in treatment for substance use disorder at an urban integrated safety-net health system. Through the use of mixed methods this study will address the following objectives: 1) To describe the family planning experiences and needs of individuals in treatment for substance use disorders (SUD) in a representative sample of patients and 2) To assess the feasibility and acceptability of the intervention among study participants. If found to be acceptable, efficacy should be assessed in a randomized controlled trial. A navigator model such as this is generalizable and could be easily integrated into a variety of settings.

ELIGIBILITY:
Inclusion Criteria:

* In treatment for substance use disorder at one of the participating clinics; 18-44 years of age; English-speaking; not currently pregnant; able to become pregnant (e.g., no history of hysterectomy, tubal ligation, hysterectomy, menopause); not planning to leave the Denver area in the next 3 months.

Exclusion Criteria:

* currently pregnant; intoxicated or mentally impaired to the point that one is unable to voluntarily consent to participate and/or respond to the surveys.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Intervention sessions completed. | up to 3 months
  Intervention acceptability will be measured by the number of sessions completed by the health educator among participants enrolled in the study.
Self-reported satisfaction with intervention. | up to 3 months
  Intervention acceptability will be assessed by participant self-reported satisfaction with the intervention (via surveys) among those who complete the intervention sessions. Satisfaction will be assessed with 8 items on a 4-point scale describing how strongly participants agree with each statement. The response scale is coded so that a higher score reflects higher satisfaction and therefore a better outcome. Reported as mean overall score (range 1-32).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Rinehart, PhD, MA, Principal Investigator — Denver Health & Hospital Authority
Locations (1):
- Denver Health & Hospital Authority, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided